CLINICAL TRIAL: NCT05182684
Title: A Multi-center Clinical Trial to Explore the Status of Collection and Transmission of Electrocardiogram Using a Wearable Device
Brief Title: The Collection and Transmission of Electrocardiogram Using a Wearable Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, SeungHwan Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VP-100-ECG
Record Dates: First submitted 2021-10-25; First posted 2022-01-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Electrocardiograms were measured by VP-100 for more than 6 hours and transmitted to a central server.
  Interventions: Device: Vital Patch(TriBell Lab)

INTERVENTIONS:
Device: Vital Patch(TriBell Lab) — Electrocardiograms were recorded using VP-100 for more than six hours and transmitted to a central data server located in Seoul National University Hospital.
  The data on a central server was confirmed and evaluated.

SUMMARY:
A multi-center clinical trial to explore the status of collection and transmission of electrocardiogram using a wearable device

DETAILED DESCRIPTION:
The collection and transmission of electrocardiograms to a central data server using a wearable device were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male volunteers who can use an Android smartphone.
* The subjects who voluntarily agree to participate and give written informed consent.

Exclusion Criteria:

* The subjects who have hypersensitivity to adhesives, such as medical bandages, or have clinically significant skin lesions.
* The subjects who are judged to be inappropriate for the clinical trials to participate.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-10-26 (Actual); Primary Completion 2022-06-21 (Estimated); Study Completion 2022-06-21 (Estimated)

PRIMARY OUTCOMES:
The proportion of data collected | 6 hours
  Compare actual monitored and server collected times

SECONDARY OUTCOMES:
The comparison of ventricular rate | 6 hours
  Compare actual monitored and server collected ventricular rate
The comparison of abnormal events | 6 hours
  Compare patient-reported adverse events with abnormal beats collected by a central server

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Seoul National University Hospital Clinical Trial Center, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huh KY, Jeong SI, Yoo H, Piao M, Ryu H, Kim H, Yoon YR, Seong SJ, Lee S, Kim KH. Lessons from a multicenter clinical trial with an approved wearable electrocardiogram: issues and practical considerations. Transl Clin Pharmacol. 2022 Jun;30(2):87-98. doi: 10.12793/tcp.2022.30.e7. Epub 2022 May 24. PMID 35800668